CLINICAL TRIAL: NCT05050435
Title: Early Cardiac Extubation After Cardiac Surgery: a Retrospective Single-center Non-inferiority Trial
Brief Title: Early Cardiac Extubation After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of department, University of Liege
Other Study IDs: Ulganescardio001
Record Dates: First submitted 2021-08-30; First posted 2021-09-20 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Post-operative Cardiac Surgery
Keywords: post-operative complications; on table extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early extubated (in operating room) patients after valvular cardiac surgery
  Interventions: Procedure: Early extubation
- Later extubated (in ICU) patients after valvular cardiac surgery

INTERVENTIONS:
Procedure: Early extubation — Patients of the 2 groups are extubated at different moments: either immediately postoperatively, in the operating room, or after a few hours monitoring in ICU
  Groups: Early extubated (in operating room) patients after valvular cardiac surgery

SUMMARY:
The management of heart valve disease is constantly evolving over time. The minimally invasive approach (mini-thoracotomy and J-hemisternotomy) is one of the major surgical evolutions. It has many advantages including, among others, a reduction of postoperative pain and the preservation of sternal stability This evolution of the surgical technique towards a less invasive approach encouraged the investigators to adapt the anesthetic management accordingly. In particular, immediate postoperative extubation appeared feasible. The investigators would therefore like to test the hypothesis that immediate extuation is non-inferior to delayed extubation with regard to patient safety. The investigators also investigated whether immediate extubation could be beneficiel in terms of vasopressors requirement, risk of early postoperative complications, fluid balance and length of stay in the intesive care unit and in the hopsital.

ELIGIBILITY:
Inclusion Criteria:

* Minimally invasive valve replacement intervention (thoracotomy or J-hemisternotomy)

Exclusion Criteria:

* Combined surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included all the patients who have had minimally invasive valve replacement surgery in our service
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications | 30 days
  Intensive care unit length of stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- ULiege - CHU, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided